CLINICAL TRIAL: NCT01723137
Title: Measuring Changes in Acute Pain in the Emergency Department Using Patient Reported Scales
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 10-3189
Record Dates: First submitted 2012-10-31; First posted 2012-11-07 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Acute Pain
Keywords: Pain; Pain measurement; Visual analog scale; Anxiety; Stress; Opioid; Emergency department; Demographics
MeSH Terms: conditions — Acute Pain; Pain; Anxiety Disorders; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- In pain: Patients who report pain greater than or equal to 3 out of 10 are eligible for this study.

SUMMARY:
Patient reported pain, stress, and anxiety measures have been found to be inter-related, but it is not known if they are all associated with receiving opiate medications. The objective of this study is to determine if patients' degree of reported pain, stress, or anxiety is associated with receiving opiate pain medications in the emergency department or at discharge. Alert patients at least 18 years of age and who report pain greater than 3/10 are eligible to participate in the study. Consenting patients complete Visual Analog Scales describing their perceived pain, stress, and anxiety from enrollment until discharge. Demographic data and administration of pain medication is also recorded. Visual Analog Scale scores among patients who received an opioid pain medicine in the emergency department and at discharge will be compared to those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Reported pain greater than or equal to 3 out of 10

Exclusion Criteria:

* Less than 18 years of age
* Decreased level of consciousness
* Inability to answer questions
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department at an urban county hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3630 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Described Stress | Immediately upon enrollment, every 30 minutes after until hospital discharge, and upon discharge, for up to 24 hours.
  Patients describe stress by completion of 100 mm Visual Analog Scale, bordered by the words "no stress" and "most stress possible".
Change in Patient described anxiety. | Immediately upon study enrollment, every 30 minutes post-enrollment, and upon hospital discharge, for up to 24 hours.
  Patients describe anxiety by completing 100mm Visual Analog Scale, bordered by the words "no anxiety" and "most anxiety possible".
Change in patient described satisfaction with ongoing treatment. | Immeditately upon enrollment, every 30 minutes post-enrollment, and upon hospital discharge, up to 24 hours.
  Patients describe satisfaction with ongoing treatment by completion of 100mm Visual Analog Scale, bordered by the words "not satisfied at all" and "completely satisfied".
Change in patient described pain. | Immediately upon enrollment, every 30 minutes post-enrollment, and upon discharge, for up to 24 hours.
  Patients describe pain by completing a 100mm Visual Analog Scale, bordered by the words "no pain" and "worst pain possible".

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States